CLINICAL TRIAL: NCT02875132
Title: An Open-label Phase II Study of Pembrolizumab in East Asian Patients With Advanced/Metastatic Acral Lentiginous Melanoma
Brief Title: Pembrolizumab in Advanced/Metastatic Acral Lentiginous Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CCTU, Comprehensive Clinical Trial Unit, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEL001
Record Dates: First submitted 2016-08-07; First posted 2016-08-23 (Estimated); Results first posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Acral Lentiginous Melanoma
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pembrolizumab (Experimental)
  Interventions: Drug: pembrolizumab

INTERVENTIONS:
Drug: pembrolizumab — pembrolizumab at 200mg IV infusion every 3 weeks

SUMMARY:
To determine the Overall Response Rate (ORR), as defined as rate of complete response (CR) and partial response (PR) as per RECIST 1.1 in biological treatment-naïve patients with acral lentiginous melanoma treated with pembrolizumab

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial.
* Be 18 years of age on day of signing informed consent.
* Have measurable disease based on RECIST 1.1.
* Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the Sponsor.
* Have a performance status of 0 or 1 on the ECOG Performance Scale.
* Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 10 days of treatment initiation.
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for more than 1 year.
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known history of active TB (Bacillus Tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., equal and less than Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., equal and less than Grade 1 or at baseline) from adverse events due to a previously administered agent.

  * Note: Subjects with equal and less than Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
  * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least eight weeks prior to the first dose of trial treatment), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Oncology, Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pembrolizumab
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Hong Kong | 9

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Overall Response Rate (ORR) is defined as rate of complete response (CR) and partial response (PR) as per RECIST 1.1 in biological treatment-naïve patients with acral lentiginous melanoma treated with pembrolizumab
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 9
participants | 1 [0 to 31.6]

2. Secondary Outcome: Response Duration
Time Frame: 2 years
Measure: Number; unit: months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 1
months | 19

3. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: To determine the Clinical Benefit Rate (CBR) of pembrolizumab treatment naïve acral lentiginous melanoma patients as defined by rate of CR + PR and stable disease (SD) of >/= 6 months
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 9
Participants | 4

4. Secondary Outcome: Progression-free Survival (PFS)
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 9
months | 3.4 [1.4 to 21.3]

5. Secondary Outcome: Overall Survival (OS)
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 9
months | 7.6 [2 to 34.3]

6. Secondary Outcome: Response Assessment as Per the Immune-related Response Criteria (irRC)
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 9
Participants | 0

7. Secondary Outcome: Number of Participants With Adverse Events
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 9
participants | 2

ADVERSE EVENTS:
Time Frame: Through study completion, up to 35 months.
Description: Number of Participants at Risk: 9
Arm/Group | Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 4/9
Serious Adverse Events (participants affected / at risk) | 4/9
Other Adverse Events (participants affected / at risk) | 2/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=9)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dizziness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Malaise (Nervous system disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=9)
Dizziness (General disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-09): https://cdn.clinicaltrials.gov/large-docs/32/NCT02875132/Prot_SAP_000.pdf